CLINICAL TRIAL: NCT01838304
Title: A Prospective, Randomized Comparison of Depth of Sedation With Propofol Titrated by Probability Ramp Control to Control by Anesthesia Providers During Esophagogastroduodenoscopy (EGD)
Brief Title: Probability Ramp Control of Propofol for EGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 817166
Record Dates: First submitted 2013-04-12; First posted 2013-04-24 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Gastrointestinal Disease
Keywords: propofol sedation endoscopy
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monitoring (Active Comparator): Standard of care sedation by CRNA using proposal with manual recording of drug dosing
  Interventions: Device: Monitoring
- Probability ramp control (Experimental): Propofol titrated to deep sedation using PRC software.
  Interventions: Device: Probability ramp control

INTERVENTIONS:
Device: Probability ramp control — Decision support software that calculates propofol doses appropriate for age and weight of the patient
  Arms: Probability ramp control
Device: Monitoring — Manual recording of drug doses determined by CRNA
  Other Names: Manual recording of drug doses determined by CRNA
  Arms: Monitoring

SUMMARY:
Endoscopic sedation requires titration of propofol to deep sedation without minimum overshoot into general anesthesia. This skill is demanding and acquired slowly. Probability Ramp Control (PRC) simplifies this by providing the clinician with a simple infusion sequence that permits gradual titration of propofol. The purpose of this study is to compare the performance of this technology to that of experienced anesthesia providers in endoscopic sedation.

DETAILED DESCRIPTION:
Administration of propofol to achieve a target of moderate sedation is a challenging task for which anesthesia providers receive minimal training. Undersedation results in a noncompliant patient, while oversedation results in airway obstruction, respiratory depression, and hypotension. Considerable variability in patient pharmacokinetics (the distribution of drug within the body) and pharmacodynamics (the translation of drug concentration to clinical effect) has been demonstrated. The skill of titrating propofol to the desired target and maintaining this state is slowly acquired in the clinical environment of the endoscopy center with frequent reliance on rescue skills. An automated system that facilitates this process would be useful.

Pharmacokinetic models allow us to make predictions of the results of drug administration. If we know the age and size of the patient, we can determine a quantity of propofol that will attain a desired concentration at some point in the future (within the predictive accuracy of the model). If they are old, this is less than if they are young. If they are obese, this is more than if they are thin. By adjusting the dosing, we can achieve similar concentrations at a specified time in a wide range of patients.

Pharmacodynamic models allow us to relate drug concentration to a probability of response. Sensitivity is a randomly distributed variable, and the cumulative probability of response to propofol is well represented by a sigmoid curve. While we do not know the concentration that will suffice for a given individual, we can determine the probability that this individual will lose responsiveness within an interval of concentrations. For example, the probability of loss of responsiveness between 1 µg/ml and 6 µg/ml is around 99%. For any given age and size, an infusion sequence can be determined so that we traverse this interval smoothly. The infusion sequence is determined by minimization of the difference between the simulated probability and the target (1). We predict that 90% of 50 year old 70 kg patients will lose responsiveness between one minute and three minutes after initiating the infusion, and 99% by five minutes. The infusion sequence for this patient is comprised of a bolus of 287 µg/kg followed by an initial infusion of 216 µg/kg/min, with an increase to 550 µg/kg/min after 147 seconds. By selecting the infusion sequence based on the age and size of the patient, all patients will track the same target line. These infusion rates are determined prior to initiation of sedation, and the clinician can verify that they are appropriate for the patient before beginning sedation.

Once the endpoint of adequate sedation is observed, the effect site concentration associated with this endpoint is inferred, and the infusion that will maintain this concentration can be determined. This allows the clinical observation to be translated into an infusion rate, much as a driver accelerates to a desired speed and then engages the cruise control to maintain that speed.

The intent of this study is to demonstrate equivalent safety and efficacy of PRC to control by a skilled clinician.

References

1. Mandel JE, Sarraf E. The Variability of Response to Propofol Is Reduced When a Clinical Observation Is Incorporated in the Control: A Simulation Study. Anesthesia & Analgesia. 2012;114:1221-9.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective EGD

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff E Mandel, MD MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Endoscopy Center, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandel JE, Sarraf E. The variability of response to propofol is reduced when a clinical observation is incorporated in the control: a simulation study. Anesth Analg. 2012 Jun;114(6):1221-9. doi: 10.1213/ANE.0b013e31824cb853. Epub 2012 Mar 30. PMID 22467886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monitoring | Probability Ramp Control
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monitoring | Probability Ramp Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (14.2) | 52.8 (16.5) | 50.625 (15.345)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 12 | 7 | 19
ASA 3 [Count of Participants; unit: Participants] — American Society of Anesthesia physical status rating. ASA 1 = Healthy ASA 2 = Minor illness (i.e. hypertension) ASA 3 = Major illness (i.e. S/P myocardial infarction)
  Participants | 7 | 8 | 15
Weight [Mean (Standard Deviation); unit: kg] | 82.3 (27.4) | 82.1 (23.9) | 82.22 (25.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Adjustment in Propofol Dosing
Description: Following initial sedation, an infusion rate for propofol is determined by the CRNA (control) or software (experimental). If this rate is appropriate for the duration of the brief procedure, no adjustment to the rate will be required. A greater requirement for rate changes suggests that the anesthesia provider needs to be immediately available to perform these adjustments.
Time Frame: Intraprocedure (average of 9 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Monitoring | Probability Ramp Control
Number analyzed (Participants) | 19 | 20
Participants | 16 | 2

2. Secondary Outcome: Decrease in Minute Ventilation From Baseline
Description: Minute ventilation as determined by respiratory inductance plethysmography from initiation of sedation until emergence.
Time Frame: Duration of sedation (average of 25 minutes)
Measure: Median (97.5% Confidence Interval); unit: percentage of baseline
Arm/Group | Monitoring | Probability Ramp Control
Number analyzed (Participants) | 19 | 20
percentage of baseline | 25 [20 to 30] | 50 [35 to 65]

3. Secondary Outcome: Time Spent Below a Saturation of 80%
Description: Number of seconds spent below saturation of 80%, reported as the total per group
Time Frame: Duration of sedation (mean 25 minutes)
Measure: Count of Units; unit: seconds
Units Other Than Participants: seconds
Arm/Group | Monitoring | Probability Ramp Control
Number analyzed (Participants) | 20 | 20
Number analyzed (seconds) | 29686 | 30552
seconds | 168 | 22
Statistical Analysis 1: Comparison: Monitoring vs Probability Ramp Control; Fisher's exact test for odd's ratio of time below a saturation of 80% to total time; Test type: Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 7.9, 95% CI 2-sided [4.21 to 14.81]

4. Secondary Outcome: Procedure Time
Description: Time from endoscopic intubation until completion of the procedure. This is not really an outcome measure, but is used to assess balance between groups.
Time Frame: Procedure time (average of 9 minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Monitoring | Probability Ramp Control
Number analyzed (Participants) | 20 | 20
minutes | 9.03 (3.75) | 8.9 (4.75)

ADVERSE EVENTS:
Time Frame: Duration of sedation (mean 25 minutes)
Arm/Group | Monitoring | Probability Ramp Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monitoring (N=20) | Probability Ramp Control (N=20)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient required bag-mask ventilation due to desaturation following propofol administration.

LIMITATIONS AND CAVEATS:
Choice of processed EEG scores in power analyasis; variability of PSI scores; lack of concealed allocation, as it was deemed unethical to ask the CRNAs to deliver "sham propofol" in the experimental arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No